CLINICAL TRIAL: NCT00422032
Title: Phase II Randomized Study of Two Different Schedules of Intravenous Clofarabine in Myelodysplastic Syndrome (MDS)
Brief Title: 2 Arm Study of Clofarabine IV in MDS Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0535
Record Dates: First submitted 2007-01-11; First posted 2007-01-15 (Estimated); Results first posted 2012-07-27 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-06

CONDITIONS: Myelodysplastic Syndrome; Leukemia
Keywords: Myelodysplastic Syndrome; Leukemia; Clofarabine; MDS
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia | interventions — Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 15 mg/m^2 Clofarabine (Experimental): Lower Dose Clofarabine Group A: 15 mg/m^2 intravenous (IV) over 1 hour daily for 5 days
  Interventions: Drug: Clofarabine
- 30 mg/m^2 Clofarabine (Experimental): Higher Dose Clofarabine Group B: 30 mg/m^2 IV over 1 hour daily for 5 days
  Interventions: Drug: Clofarabine

INTERVENTIONS:
Drug: Clofarabine — Group A: 15 mg/m^2 IV over 1 hour daily for 5 days
  Group B: 30 mg/m^2 IV over 1 hour daily for 5 days
  Other Names: Clolar

SUMMARY:
The goal of this clinical research study is to compare the effectiveness of 2 different doses of the drug clofarabine that can be given on a weekly schedule for the treatment of Myelodysplastic Syndrome (MDS). The safety of these two doses will also be compared.

Primary Objective: Compare the response rates of two dose schedules of clofarabine in MDS.

Secondary Objective: Compare response durations, survivals and side effects of the two schedules.

DETAILED DESCRIPTION:
Clofarabine is a new chemotherapy drug that is designed to interfere with the growth and development of cancer cells.

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the toss of a coin) to one of two treatment groups (Groups A and B). Participants in Group A will receive a lower dose of clofarabine. Participants in Group B will receive a higher dose of clofarabine. At first, there will be an equal chance of being assigned to either group. However, as experience increases and more information becomes available, the chance of being assigned to the group that has shown the most effectiveness will increase. You and the study doctor will know to which group you are assigned.

Participants will receive clofarabine as a 1-hour infusion into a vein once a day for 5 days in a row. This will be repeated every 4 to 8 weeks. Each 4-8 week period is considered 1 cycle of treatment.

For participants in both groups, after each cycle of therapy, they will not receive the next cycle of chemotherapy until their blood counts have recovered and any possible side effects have gone away (for around 4 to 8 weeks). You must stay in Houston for the first treatment cycle (about 4 to 8 weeks) and will be required to return to Houston before receiving each additional cycle of chemotherapy (up to 6 days each cycle).

Before every treatment cycle, your doctor will perform a physical exam, including measurement of your weight and vital signs (blood pressure, heart rate, temperature, and breathing rate). You will be asked about the level of your daily activities and how you are feeling. You will have blood samples (about 1-2 teaspoons) collected for routine lab tests 1-2 times a week for the first cycle, then every 2-4 weeks while on therapy. Repeat bone marrow samples will be collected every 1-3 cycles. However, if you complete the study before the third cycle, the bone marrow may be taken then. You may choose to have check-up visits and blood tests with your local doctor.

If you show a response and do not experience any severe side effects, you can receive up to a total of 12 cycles of therapy. During each cycle, clofarabine will be given the same way as during the first cycle. However, the dose of clofarabine may be lowered during later cycles to decrease the risk of side effects that may have occurred in previous cycles. If the disease gets worse or you experience any intolerable side effects, you will be taken off the study and your doctor will discuss other treatment options with you.

This is an investigational study. Clofarabine is approved by the FDA for treatment of pediatric acute lymphoblastic leukemia. Its use in this study is experimental. Up to 60 participants will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with MDS and >/= 5% blasts or International Prognostic Scoring System (IPSS) risk intermediate or high; patients with Chronic Myelomonocytic Leukemia (CMML).
2. No prior intensive chemotherapy or high-dose ara-C (> 1g/m2).
3. Prior biologic therapies, targeted therapies, or single agent chemotherapy allowed.
4. Patients must have been off chemotherapy for 2 weeks prior to entering this study and recovered from the toxic effects of that therapy, unless there is evidence of rapidly progressive disease.
5. Hydroxyurea is permitted for control of counts prior to treatment.
6. Procrit, GCSF are allowed before therapy.
7. Performance 0-2 (Eastern Cooperative Oncology Group (ECOG)). Adequate organ function including the following: Adequate liver function (bilirubin of < 2mg/dl), and renal function (creatinine < 2mg/dl), and SGPT (ALT) < 3 * upper limit of normal (ULN). Adequate cardiac functions (New York Heart Association (NYHA) cardiac III-IV excluded).
8. Signed informed consent.

Exclusion Criteria:

1. Nursing and pregnant females. Patients of childbearing potential should practice effective methods of contraception. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
2. Active and uncontrolled infections.
3. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements.
4. Prior clofarabine treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hagop Kantarjian, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson's Website — http://mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period 1/31/06 - 9/21/09. All patients were registered at The University of Texas M.D. Anderson Cancer Center.
Pre-assignment Details: Of the 60 participants registered on this study, two (2) were excluded prior to receiving treatment.
Period: Overall Study
Arm/Group | 15 mg/m^2 Clofarabine | 30 mg/m^2 Clofarabine
Started | 37 | 21
Completed | 37 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 15 mg/m^2 Clofarabine | 30 mg/m^2 Clofarabine | Total
Number analyzed (Participants) | 37 | 21 | 58
Age Continuous [Median (Full Range); unit: Years] | 68 [25 to 89] | 65 [34 to 83] | 68 [25 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 7 | 20
  Male | 24 | 14 | 38
Region of Enrollment [Number; unit: participants]
  United States | 37 | 21 | 58

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Response for Two Dose Schedules of Clofarabine
Description: Response defined as Complete Remission (CR): Normalization of blood counts with neutrophils >/= 1 * 10^9/L and platelet counts >/= 100 * 10^9/L, and marrow blasts </=5%; Partial Remission: as above except for presence of 6-15% marrow blasts, or 50% reduction if <15% at start of treatment; or Hematologic Improvement (HI): Complete Response (CR) with the exception of a lack of platelet recovery to >/= 100 * 10^9/L. Repeat bone marrow samples collected every 1-3 cycles (4-8 week cycle).
Time Frame: 4 weeks (minimum 1 cycle) up to 24 weeks (maximum 3 cycles of 8 weeks)
Measure: Number; unit: Participants
Arm/Group | 15 mg/m^2 Clofarabine | 30 mg/m^2 Clofarabine
Number analyzed (Participants) | 37 | 21
Participants
  Complete Response | 10 | 5
  Hematologic Improvement | 5 | 1

ADVERSE EVENTS:
Time Frame: 4 years, 10 months.
Arm/Group | 15 mg/m^2 Clofarabine | 30 mg/m^2 Clofarabine
Serious Adverse Events (participants affected / at risk) | 7/37 | 8/21
Other Adverse Events (participants affected / at risk) | 35/37 | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 15 mg/m^2 Clofarabine (N=37) | 30 mg/m^2 Clofarabine (N=21)
Acute Renal Failure (Renal and urinary disorders) | 2 (2) | 1 (1)
Hemorhage (Nervous system disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 2 (2) | 5 (5)
Febrile Neutropenia (Infections and infestations) | 1 (1) | 0 (0)
Death (General disorders) | 2 (2) | 1 (1)
Thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 15 mg/m^2 Clofarabine (N=37) | 30 mg/m^2 Clofarabine (N=21)
Nausea (Gastrointestinal disorders) | 23 (23) | 13 (13)
Skin Rash (Skin and subcutaneous tissue disorders) | 16 (16) | 8 (8)
Transaminase elevations (Metabolism and nutrition disorders) | 13 (13) | 14 (14)
Diarrhea (Gastrointestinal disorders) | 10 (10) | 6 (6)
Vomiting (Gastrointestinal disorders) | 9 (9) | 8 (8)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 7 (7) | 6 (6)
Headache (Nervous system disorders) | 5 (5) | 4 (4)
Elevated Creatinine (Metabolism and nutrition disorders) | 2 (2) | 6 (6)
Mucositis (Gastrointestinal disorders) | 4 (4) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Myalgia/bone pain (General disorders) | 2 (2) | 2 (2)
Fatigue (General disorders) | 2 (2) | 1 (1)
Edema (General disorders) | 2 (2) | 1 (1)
Acute Renal Failure (Renal and urinary disorders) | 0 (0) | 3 (3)
Congestive Heart Failure (Cardiac disorders) | 0 (0) | 1 (1)
Weakness (General disorders) | 0 (0) | 1 (1)
Prolonged Myelosuppression (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No